CLINICAL TRIAL: NCT03802214
Title: A Case-control Study to Evaluate the Immunoinflammatory Effect of Prior Exposure to Anti-TNF Therapy in Patients With Ulcerative Colitis Starting Vedolizumab Therapy
Brief Title: Ulcerative Colitis - Vedolizumab- With/Without Prior Exposure to Anti-TNF（Tumor Necrosis Factor）Therapy
Status: Terminated | Type: Observational
Why Stopped: Funding discontinued
Sponsor: Stanford University (Other)
Collaborators: Takeda (Industry); University of Western Ontario, Canada (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Aida Habtezion, Associate Professor, Stanford University
Other Study IDs: IRB48889
Record Dates: First submitted 2018-12-10; First posted 2019-01-14 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — collection of blood and tissue specimens for immunology and drug assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- vedolizumab-UC-naïve to TNF-antagonist: standard vedolizumab induction therapy for ulcerative colitis patients who are naïve to TNF-antagonist therapy
  Interventions: Drug: Vedolizumab
- vedolizumab-UC- previous TNF-antagonist: standard vedolizumab induction therapy for ulcerative colitis patients with previous TNF-antagonist exposure
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — standard vedolizumab induction (300mg IV at week 0, 2, 6)
  Other Names: Entyvio

SUMMARY:
A case-control study to evaluate the immunoinflammatory effect of prior exposure to anti-TNF therapy in patients with ulcerative colitis starting vedolizumab therapy

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD)- ulcerative colitis (UC) and Crohn's disease (CD)- are chronic conditions of the gastrointestinal tract. Treatment generally consists of immunosuppression to modify the dysregulated immune responses. Vedolizumab, an inhibitor of α4β7, is a highly effective therapy for treating IBD, that minimized adverse effects through its gut selective inhibition of lymphocyte trafficking. However, the mechanism of action remains incompletely characterized especially in those previously treated to other biologics and why some patients are either vedolizumab non-responders or fail to respond over time. We would like to address the question whether anti-TNF non-responders as well as those that either do not respond or fail overtime to respond to vedolizumab identifies a specific population with difficult to treat disease that have alternate trafficking patterns and whether prior exposure to anti-TNF alters the mucosal immune responses, and/or trafficking patterns when compared to anti-TNF naive patients that may help explain impaired response to vedolizumab induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years old)
* clinical diagnosis of inflammatory bowel disease (Ulcerative Colitis)
* clinical indication for biologic therapy
* naive or failed anti-TNF therapy previously

Exclusion Criteria:

* patients allergic or intolerant to vedolizumab,
* past use of vedolizumab;
* patient unable to give consent to enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical indication for biologic therapy, adult patients (>18) with the diagnosis of inflammatory bowel disease (Ulcerative Colitis) who are naive or failed anti-TNF therapy previously.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Analysis of blood and tissue leukocytes (T cells, B cells and Dendritic cells) | changes from enrollment to end of treatment (week 14)
  Analysis of blood and tissue leukocytes (T cells, B cells and Dendritic cells) in patients with and without prior anti-TNF exposure

SECONDARY OUTCOMES:
Analysis of the serum and tissue concentrations of inflammatory markers (interleukins) | changes from enrollment to end of treatment (week 14)
  Analysis of the serum and tissue concentrations of inflammatory markers (interleukins) in vedolizumab responders versus non-responders
Analysis of the serum and tissue concentrations of vedolizumab | changes from enrollment to end of treatment (week 14)
  Analysis of the serum and tissue concentrations of vedolizumab in patients with and without prior anti-TNF exposure

CONTACTS AND LOCATIONS:
Overall Officials: Aida Habtezion, MD, Principal Investigator — Stanford University
Locations (2):
- Stanford University, Stanford, California, United States
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We will share the data through the publication of results. Individual participant data was not promised to be shared.

REFERENCES:
- [Background] Schmitt H, Billmeier U, Dieterich W, Rath T, Sonnewald S, Reid S, Hirschmann S, Hildner K, Waldner MJ, Mudter J, Hartmann A, Grutzmann R, Neufert C, Munster T, Neurath MF, Atreya R. Expansion of IL-23 receptor bearing TNFR2+ T cells is associated with molecular resistance to anti-TNF therapy in Crohn's disease. Gut. 2019 May;68(5):814-828. doi: 10.1136/gutjnl-2017-315671. Epub 2018 May 30. PMID 29848778
- [Background] Boden EK, Shows DM, Chiorean MV, Lord JD. Identification of Candidate Biomarkers Associated with Response to Vedolizumab in Inflammatory Bowel Disease. Dig Dis Sci. 2018 Sep;63(9):2419-2429. doi: 10.1007/s10620-018-4924-8. Epub 2018 Jan 25. PMID 29372476
- [Background] Suzawa K, Kobayashi M, Sakai Y, Hoshino H, Watanabe M, Harada O, Ohtani H, Fukuda M, Nakayama J. Preferential induction of peripheral lymph node addressin on high endothelial venule-like vessels in the active phase of ulcerative colitis. Am J Gastroenterol. 2007 Jul;102(7):1499-509. doi: 10.1111/j.1572-0241.2007.01189.x. Epub 2007 Apr 24. PMID 17459027
- [Background] Kobayashi M, Hoshino H, Masumoto J, Fukushima M, Suzawa K, Kageyama S, Suzuki M, Ohtani H, Fukuda M, Nakayama J. GlcNAc6ST-1-mediated decoration of MAdCAM-1 protein with L-selectin ligand carbohydrates directs disease activity of ulcerative colitis. Inflamm Bowel Dis. 2009 May;15(5):697-706. doi: 10.1002/ibd.20827. PMID 19067429
- [Background] Sandborn WJ, Feagan BG, Rutgeerts P, Hanauer S, Colombel JF, Sands BE, Lukas M, Fedorak RN, Lee S, Bressler B, Fox I, Rosario M, Sankoh S, Xu J, Stephens K, Milch C, Parikh A; GEMINI 2 Study Group. Vedolizumab as induction and maintenance therapy for Crohn's disease. N Engl J Med. 2013 Aug 22;369(8):711-21. doi: 10.1056/NEJMoa1215739. PMID 23964933
- [Background] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, Van Assche G, Axler J, Kim HJ, Danese S, Fox I, Milch C, Sankoh S, Wyant T, Xu J, Parikh A; GEMINI 1 Study Group. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013 Aug 22;369(8):699-710. doi: 10.1056/NEJMoa1215734. PMID 23964932
- [Background] Rosario M, Dirks NL, Gastonguay MR, Fasanmade AA, Wyant T, Parikh A, Sandborn WJ, Feagan BG, Reinisch W, Fox I. Population pharmacokinetics-pharmacodynamics of vedolizumab in patients with ulcerative colitis and Crohn's disease. Aliment Pharmacol Ther. 2015 Jul;42(2):188-202. doi: 10.1111/apt.13243. Epub 2015 May 20. PMID 25996351